CLINICAL TRIAL: NCT06209554
Title: The Efficacy of Diode Laser and Subgingival Air Polishing With Erythritol in Treatment of Periodontitis ( Clinical and Microbiological Study)
Brief Title: The Efficacy of Diode Laser and Subgingival Air Polishing With Erythritol in Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: sara mohamed awad elmeligy (Other)
Responsible Party: Sponsor-Investigator, sara mohamed awad elmeligy, Investigator Affiliation, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: treatment of periodontitis
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Periodontitis
Keywords: Diode laser, Erythritol
MeSH Terms: conditions — Periodontitis | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Experimental): Eight patients to be treated with only Scaling and root planning .
  Interventions: Device: ultrasonic tips and Gracey curettes, airflow with erythritol and diode laser
- erythritol group (Experimental): Eight patients to be treated with erythritol air polishing as an adjunct to Scaling and root planning .
  Interventions: Device: ultrasonic tips and Gracey curettes, airflow with erythritol and diode laser
- laser group (Experimental): Eight patients to be treated with dioad laser as an adjunct to Scaling and root planning .
  Interventions: Device: ultrasonic tips and Gracey curettes, airflow with erythritol and diode laser

INTERVENTIONS:
Device: ultrasonic tips and Gracey curettes, airflow with erythritol and diode laser — diode laser and erythritol used as adjunctive method in the treatment of periodontitis in addition to scaling and root planning

SUMMARY:
The present study aims to evaluate the efficacy of subgingival air polishing by erythritol and diode laser in the treatment of periodontitis (clinically and microbiologically).

DETAILED DESCRIPTION:
Periodontitis, a chronic condition, leads to inflammation of the periodontium, resulting in the degradation of the periodontal ligament and adjacent alveolar bone, potentially leading to tooth loss The oral cavity, hosting nearly 700 distinct bacteria, is the primary origin of periodontitis, where bacterial pathogens trigger an inflammatory response, causing connective tissue deterioration. Gram-negative bacteria, including Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, and Tannerella forsythia, contribute to periodontitis.

Dental plaque illustrates bacterial growth in the form of a biofilm Porphyromonas gingivalis, a Gram-negative anaerobic bacterium, is found in 85.75% of subgingival plaques associated with chronic periodontitis. The presence of Aggregatibacter actinomycetemcomitans at the individual level is notably associated with disease risk due to its genetic variation and virulence factors.

Exclusive reliance on mechanical therapy (SRP) may fall short in eliminating pathogenic bacterial species due to their presence within periodontal tissues or in regions inaccessible by periodontal instruments during close debridement. These challenges pose constraints on the enduring stability of outcomes in nonsurgical techniques, forming the rationale for supplementary therapies involving antibiotics, antiseptics, nonchemical modalities, laser, and photodynamic therapy.

Laser therapy, particularly the diode laser at 940 nm, in conjunction with SRP, enhances and facilitates the healing process in treated sites. The diode laser, preferred for its cost-effectiveness, portability, and user-friendly nature, simultaneously addresses the removal of diseased soft tissues, targets microorganisms, and induces an antibacterial effect within periodontal pockets.

Its favorable tissue penetration capabilities and absorption in pigmented tissues make it particularly adept at targeting pigmented bacteria and granulation tissue.

The emergence of low-abrasive and resorbable powders, used with subgingival delivery tools, sparks renewed interest in air-polishing devices (APDs) for periodontal treatment. Research indicates that APDs contribute to a reduction in post-operative patient discomfort and sensitivity, enhance patient acceptance, and result in minimal alterations to surrounding soft and hard tissues. Air-flow therapy may be particularly beneficial for challenging cases such as teeth with furcation involvement and sites with restricted access, traditionally posing difficulties for thorough debridement using conventional instrumentation.

Initially designed to eliminate biofilm and stains, APDs using abrasive powders were found detrimental to exposed root surfaces, gingiva, and certain restorative materials. Subsequently, there was a shift towards the adoption of resorbable powders with low abrasiveness, including glycine and erythritol, to mitigate adverse effects.

The recently introduced erythritol powder, a water-soluble, non-toxic sugar alcohol, and artificial sweetener, is extensively employed in the food industry. Erythritol powder air-polishing (EPAP) used as a monotherapy exhibits outcomes in supportive periodontal therapy comparable to those achieved through conventional power-driven and manual debridement.

There is a suggestion that erythritol powder may possess a prolonged antimicrobial effect on the subgingival biofilm, with studies indicating its capability to decrease the numbers of P. gingivalis and Aggregatibacter actinomycetemcomitans during supportive periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients. Patient with stageІ& stage ІІ periodontitis according to Classification of periodontal and peri-implant diseases and conditions 2017

Exclusion Criteria:

* Patients with any systemic disease linked to delayed wound healing, such as uncontrolled diabetes, autoimmune diseases, heart conditions, etc.

Current smokers. Patients underwent prior periodontal therapy within the last 6 months. Individuals who had used antibiotics in the previous 6 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
probing depth and clinical attachment loss | baseline and 6 weeks follow up
  decreasing probing depth and clinical attachment loss refer to healing of periodontal pocket

CONTACTS AND LOCATIONS:
Overall Officials: samah H elmeadawy, ph.D, Study Chair — Mansoura U
Locations (1):
- Mansoura Univeristy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
it is difficult to be in direct contact with patient after work is finished ,due to the distance.

REFERENCES:
- [Derived] Elmeligy SMA, Saleh W, Elewa GM, Abu El-Ezz HZ, Mahmoud NM, Elmeadawy S. The efficacy of diode laser and subgingival air polishing with erythritol in treatment of periodontitis (clinical and microbiological study). BMC Oral Health. 2024 Jul 4;24(1):763. doi: 10.1186/s12903-024-04481-6. PMID 38965550